CLINICAL TRIAL: NCT02019953
Title: Effects of Health-Promoting Programs on Cardiovascular Disease Risk: JHS
Brief Title: Effects of Health Promoting Programs on Cardiovascular Disease Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Gailen D. Marshall Jr., MD PhD, Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2010-0057
Record Dates: First submitted 2013-04-30; First posted 2013-12-24 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Yoga; Walking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Yoga 3 times per week (Other): Yoga participation 3 x per week for 24 weeks; 48 week follow-up.
  Interventions: Other: Yoga
- Yoga 2 times per week (Other): Yoga participation 2 x per week for 24 weeks; 48 week follow-up
  Interventions: Other: Yoga
- Yoga 1 time per week (Other): Yoga participation 1 x per week for 24 weeks; 48 week follow-up
  Interventions: Other: Yoga
- Walking 3 times per week (Other): Walking 3x per week for 24 weeks; 48 week follow-up
  Interventions: Other: Walking
- Healthy Lifestyles Education (Other): Healthy Lifestyles Education Participation 1 x per week for 24 weeks; 48 week follow-up
  Interventions: Other: Healthy Lifestyles Education

INTERVENTIONS:
Other: Yoga — The yoga intervention, which is taught based on Hatha yoga, will be offered to study participants in Study Arms 1, 2, and 3, is a combination of asanas (poses), pranayams (breathing exercises), and meditation. Blood pressure and heart rate measurements are taken before and after each session.
  Arms: Yoga 1 time per week; Yoga 2 times per week; Yoga 3 times per week
Other: Walking — The walking intervention, which is Study Arm 4 includes, three guided walking sessions per week for 24 weeks. Each class is an hour in length and will include a minimum of 30 minutes of walking at the equivalent of a minimum of three miles per hour. Each session includes a ten-minute warm-up and ten-minute cool-down period of some stretches and walking at a leisurely pace. Blood pressure and heart rate measurements are taken before and after each session.
  Arms: Walking 3 times per week
Other: Healthy Lifestyles Education — Participants randomly assigned to the fifth study arm attend one 60-minute healthy lifestyles class per week for 24 weeks. The Healthy Lifestyles curriculum includes 24 independent lesson modules, which allows participants to begin their intervention at any time during the course schedule. Blood pressure and heart rate measurements are taken before and after each session.
  Other Names: Health Education
  Arms: Healthy Lifestyles Education

SUMMARY:
The overall approach to the study is to assess the feasibility of recruiting African Americans to participate in several health-promoting programs and to compare health outcomes among the three interventions.

DETAILED DESCRIPTION:
The project is designed to achieve five specific aims: (1) To determine the feasibility of attracting African Americans into Health Promotion Research studies;(2) To determine whether clinically recorded information can be used as a guide for recruitment inclusion in Health Promotion Studies from an active epidemiological research cohort;(3) To measure the ability to retain African Americans recruited into Health Promotion Studies from an active research cohort;(4) To measure the adherence to various protocols within a Health promotion Study; and(5) To provide informed estimates of effect sizes for designing future Health Promotion Research.

A total of 375 study participants from the Jackson Heart Study (JHS) cohort, all of whom are African American, will be randomly assigned to one of five, equally-sized study arms: (1) practicing yoga three times per week; (2) practicing yoga two times per week; (3) practicing yoga one time per week; (4) walking briskly three times per week; and (5) attending a weekly healthy lifestyles class.

All study arms will include a 24-week intervention. In addition, participants will have a total of four clinical visits with members of the study team baseline, 12 weeks, 24 weeks, and 48 weeks) in which the following measures will be recorded:

1. Systolic and diastolic blood pressure and heart rates
2. Highly sensitive C-reactive protein (hsCRP) - serum, fibrinogen - plasma (sodium citrate), homocysteine (plasma), and interleukin-6 levels (IL-6) (serum).
3. Fasting total cholesterol, low density (LDL), direct high density lipoprotein (HDL), and triglyceride levels - all serum
4. HbA1c level
5. BMI, waist circumference
6. Medication and supplement use and dosages
7. Results of a study survey designed to measure participants' changes in their reported health-related quality of life, perceived stress, health behaviors, sleep patterns, and impact of pain on everyday life

In addition, we will also record systolic and diastolic blood pressure and heart rates before and after each intervention session for all five study arms.

ELIGIBILITY:
Inclusion Criteria:

* This study includes only one inclusion criterion: to participate in this study, one needs to be a member of the Jackson Heart Study cohort.

Exclusion Criteria:

* 1. Newly diagnosed (within the last six weeks) with a myocardial infarction, cerebrovascular disease, atrial fibrillation, cardiomyopathy, valvular heart disease, fatal cardiac arrhythmia, severe systolic and diastolic heart failure, uncontrolled COPD, uncontrolled moderate to severe hypertension, or a recent recipient of a pacemaker, and/or

  2. Change in blood pressure medicine or lipid-lowering medication up to 30 days prior to or plans for a change in the 30 days after enrollment in the study, and/or

  3. Already practicing yoga at least once per week or walking briskly for one hour at least three times per week, and/or

  4. Inability to attend protocol sessions, and/or

  5. Diagnosis of an underlying medical illness that might be considered by the principal investigator to potentially impair one's safety or ability to complete the study protocol (example could possibly include uncontrolled asthma), and/or

  6. Current use of a prescription regimen that might be considered by the principal investigator to potentially impair one's safety or ability to complete the study protocol (examples could possibly include use of sedatives or other drugs that could affect a participant's ability to participate in any of the study arms).

  7. Pregnant or planning to become pregnant in the next six (6) months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2012-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Primary outcomes for this feasibility study will focus on composite measures for recruitment, retention, and the reasons for refusal or dropout. | Bi-annual for up to 52 weeks after enrollment
  Primary outcomes for this feasibility study will focus on measures for recruitment, retention, and the reasons for refusal or dropout, and consist of (1) agreement to participate in the study (recruitment); (2) reasons for participating/not-participating; (3) dropout, defined as a monotone missingness pattern of stopping participation before completion of the study; (4) reasons for discontinuation/dropout; (5) attendance, defined as the potentially non-monotone pattern of coming to the scheduled study session; and (6) adherence, defined as attending and completing the scheduled sessions and clinical visits.

SECONDARY OUTCOMES:
Changes in participants' hypertension profiles. | 48 weeks
  Defined using measures of their systolic and diastolic blood pressure
Changes in participants' inflammation markers | 48 weeks
  Defined using measures of participants' hsCRP, fibrinogen, homocysteine, and interleukin-6 levels.
Changes in participants' lipids profiles. | 48 weeks
  Defined as using measures of participants' fasting total cholesterol, LDL, HDL, and triglycerides.
Changes in participants' HbA1c levels. | 48 weeks
  Changes in participants' HbA1c levels.
Changes in participants' reported health-related quality of life. | 48 weeks
  Quality of life measured as measured by perceived stress, health behaviors, sleep patterns, and impact of pain on everyday life.

CONTACTS AND LOCATIONS:
Overall Officials: Gailen D Marshall, MD, PhD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No